CLINICAL TRIAL: NCT06946602
Title: Bu/Cy/Flu/ATG Versus Bu/Cy/ATG Conditioning Regimen in Elderly AML Patients Receiving Haploidentical Hematopoietic Stem Cell Transplantation: a Prospective, Randomized, Controlled Study
Brief Title: Conditioning Regimen in Elderly AML Patients Receiving Haplo-HSCT.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Sun Yuqian, Associate Professor, Peking University People's Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025PHB096-001; Peking University (Registry Identifier: Peking University)
Record Dates: First submitted 2025-04-19; First posted 2025-04-27 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: AML; Elderly
Keywords: Haplo-HSCT; elderly; AML; RIC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bu/Flu/Cy/ATG (Experimental)
  Interventions: Procedure: Bu/Flu/Cy/ATG
- Bu/Cy/ATG (Active Comparator)
  Interventions: Procedure: Bu/Cy/ATG

INTERVENTIONS:
Procedure: Bu/Flu/Cy/ATG — The Bu/Flu/Cy/ATG conditioning regimen consists of the following components: Ara-C (2 g/m²/day, injected i.v.) on days-10 and-9; Bu (0.8 mg/kg, q6h, injected i.v.) on days -8 to -6; Flu (30 mg/m²/day, injected i.v.) from day-6 to day-2; Cy (1.0 g/m²/day, injected i.v.) on days-5 and-4; and ATG (2.5 mg/kg/day) on days-5 to -2.
  Arms: Bu/Flu/Cy/ATG
Procedure: Bu/Cy/ATG — The Bu/Cy/ATG conditioning regimen consists of the following components: Ara-C (4 g/m²/day, injected i.v.) on day-9; Bu (0.8 mg/kg, q6h, injected i.v.) on days -8 to -6; Cy (1.8 g/m²/day, injected i.v.) on days-5 and-4; and ATG (2.5 mg/kg/day) on days-5 to -2.
  Arms: Bu/Cy/ATG

SUMMARY:
Elderly AML patients receiving conventional chemotherapy have poor prognosis. Allo-HSCT offers better long-term survival than chemotherapy, while high TRM limits its use. Current research focuses more on improving conditioning regimens to reduce TRM. Studies suggest Bu/Flu/Cy/ATG are safer and more effective for elderly AML haplo-HSCT, lowering TRM. However, prospective randomized trials are lacking. This study aims to compare Bu/Flu/Cy/ATG vs. Bu/Cy/ATG to determine if TRM can be reduced in elderly AML undergoing haplo-HSCT.

DETAILED DESCRIPTION:
The prognosis of elderly patients with acute myeloid leukemia (AML) undergoing conventional chemotherapy is poor. Compared with chemotherapy, allogeneic hematopoietic stem cell transplantation (allo-HSCT) can improve long-term survival in elderly patients. However, the high transplantion-related mortality (TRM) limited its application. Currently, the top priority in transplantation for elderly AML patients is to reduce TRM through methods such as optimizing conditioning regimens, reducing graft-versus-host disease (GVHD), and preventing infections. Present research primarily focuses on optimizing conditioning regimens. Both domestic and international studies, as well as our team's preliminary research, suggest that replacing cyclophosphamide (Cy) with fludarabine (Flu) can reduce toxicity. Earlier prospective single-arm clinical study in our team confirmed that the Bu/Flu/Cy/ATG regimen is a safe and effective conditioning protocol for haploidentical hematopoietic stem cell transplantation (haplo-HSCT) in elderly AML patients. This study aims to use a prospective randomized controlled trial to verify whether the Bu/Flu/Cy/ATG conditioning regimen can reduce TRM compared with the Bu/Cy/ATG regimen in elderly AML patients undergoing haplo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

- (a)Diagnosed with AML in first complete remission (CR1). (b)Age ≥55 years. (c)Availability of an haploidentical donor, first transplant, no matched sibling or unrelated donor.

(d)Willingness to provide written informed consent.

Exclusion Criteria:

* (a) Uncontrolled active infection. (b) Secondary AML. (c)Refusal to provide informed consent.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Transplant-related mortality (TRM) | From HSCT to the follow-up assessment at 12 months post-treatment.
  TRM is defined as death due to any transplantation-related cause other than disease relapse. Transplant-related mortality will be calculated using a competing risks model.

SECONDARY OUTCOMES:
Toxicity of conditioning | From HSCT to the follow-up assessment at 28 days and 100 days post-treatment.
  Toxicity of conditioning within 28 days of HSCT can be graded according to Common Terminology Criteria for Adverse Events (CTCAE): 1.Grade 1: Mild toxicity that does not require medical intervention. 2.Grade 2: Moderate toxicity that may require medical intervention. 3.Grade 3: Severe toxicity that requires significant medical intervention, hospitalization, or results in lasting effects. 4.Grade 4: Life-threatening toxicity, potentially requiring intensive care. 5.Grade 5: Death caused by the toxicity reaction.
Engraftment | Platelet engraftment was assessment at 28 days post-transplantation.
  Platelet engraftment was defined as the first of seven consecutive days with a platelet count >20 × 109/L without transfusion support. Neutrophil engraftment was defined as the first of three consecutive days with an ANC > 0.5 × 109/L.
GVHD | From HSCT to the follow-up assessment at 12 months post-treatment.
  Acute GVHD was classified as symptom presentation before 100 days after haplo-HSCT and chronic GVHD was classified as symptom presentation >100 days after haplo-HSCT. Each organ (skin, liver, and gut) was staged 1 through 4 for Acute GVHD according to modified criteria based on the schema of the Mount Sinai Acute GVHD International Consortium (MAGIC), and patients were also assigned a grade of acute GVHD (I through IV) based on overall severity. Chronic GVHD was graded in accordance with the National Institutes of Health (NIH) Chronic Graft-versus-Host Disease Consensus Criteria.
Overall Survival | From HSCT to the follow-up assessment at 12 months post-treatment.
  The time from haplo-HSCT to death from any cause in patients with AML. Overall survival will be calculated using the Kaplan-Meier method.
Cumulative Incidence of Relapse | From HSCT to the follow-up assessment at 12 months post-treatment.
  Relapse was defined as disease recurrence.
Leukemia-free survival | From HSCT to the follow-up assessment at 12 months post-treatment.
  Leukemia-free survival (LFS) was defined as the time from transplantation to relapse, disease progression, or death, whichever occurred first.
Event-Free Survival | From HSCT to the follow-up assessment at 12 months post-treatment.
  Event-Free Survival (EFS) was defined as the time from transplantation to relapse, graft failure, death from any cause, or requirement for additional anti-leukemic therapy.
Viral Infection | From HSCT to the follow-up assessment at 12 months post-treatment.
  Detection of CMV-DNA and EBV-DNA in peripheral blood twice a week.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Santoro N, Labopin M, Ciceri F, Van Lint MT, Nasso D, Blaise D, Arcese W, Tischer J, Bruno B, Ehninger G, Koc Y, Santarone S, Huang XJ, Savani BN, Mohty M, Ruggeri A, Nagler A. Impact of conditioning intensity on outcomes of haploidentical stem cell transplantation for patients with acute myeloid leukemia 45 years of age and over. Cancer. 2019 May 1;125(9):1499-1506. doi: 10.1002/cncr.31941. Epub 2019 Jan 8. PMID 30620383
- [Background] Sun YQ, Xu LP, Zhang XH, Liu DH, Chen H, Wang Y, Yan CH, Wang JZ, Wang FR, Zhang YY, Liu KY, Huang XJ. A retrospective comparison of BU-fludarabine and BU-CY regimens in elderly patients or in patients with comorbidities who received unmanipulated haploidentical hematopoietic SCT. Bone Marrow Transplant. 2015 Apr;50(4):601-3. doi: 10.1038/bmt.2014.303. Epub 2015 Jan 19. No abstract available. PMID 25599162
- [Background] Huang XJ, Zhu HH, Chang YJ, Xu LP, Liu DH, Zhang XH, Jiang B, Jiang Q, Jiang H, Chen YH, Chen H, Han W, Liu KY, Wang Y. The superiority of haploidentical related stem cell transplantation over chemotherapy alone as postremission treatment for patients with intermediate- or high-risk acute myeloid leukemia in first complete remission. Blood. 2012 Jun 7;119(23):5584-90. doi: 10.1182/blood-2011-11-389809. Epub 2012 Apr 24. PMID 22535659
- [Background] Sun YQ, Han TT, Wang Y, Yan CH, Wang FR, Wang ZD, Kong J, Chen YH, Chen H, Han W, Chen Y, Zhang YY, Zhang XH, Xu LP, Liu KY, Huang XJ. Haploidentical Stem Cell Transplantation With a Novel Conditioning Regimen in Older Patients: A Prospective Single-Arm Phase 2 Study. Front Oncol. 2021 Feb 26;11:639502. doi: 10.3389/fonc.2021.639502. eCollection 2021. PMID 33718234